CLINICAL TRIAL: NCT04292535
Title: Placebo Controlled Phase II Clinical Trial: Safety and Efficacy of Combining Intranasal Insulin & Acute Exercise
Brief Title: Safety and Efficacy of Combining Intranasal Insulin & Acute Exercise
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Matthew B. Pontifex, Ph.D., Associate Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00000804
Record Dates: First submitted 2020-02-28; First posted 2020-03-03 (Actual); Results first posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-05

CONDITIONS: Insulin; Exercise
Keywords: Intranasal Insulin; Cognition; Exercise; Physical Activity
MeSH Terms: conditions — Insulin Resistance; Motor Activity | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Random allocation to a dose of intranasal insulin (0, 20, 40, 60, 80, 100, 120) Within each dose, random allocation to exercise or control activity.
Who Masked: Participant, Investigator
Masking Description: Double blind, placebo controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Passive Control (Active Comparator): 20 minute sedentary control period during which participants watched an emotionally neutral video.
  Interventions: Drug: Placebo into the intranasal mucosa; Drug: 20 IU NovoLog Insulin aspart into the intranasal mucosa; Drug: 40 IU NovoLog Insulin aspart into the intranasal mucosa; Drug: 60 IU NovoLog Insulin aspart into the intranasal mucosa; Drug: 80 IU NovoLog Insulin aspart into the intranasal mucosa; Drug: 100 IU NovoLog Insulin aspart into the intranasal mucosa; Drug: 120 IU NovoLog Insulin aspart into the intranasal mucosa
- Acute Exercise (Experimental): 20 minute physical activity period during which participants exercised on a treadmill at an intensity corresponding to 60-65% of maximum heart rate while watching an emotionally neutral video.
  Interventions: Drug: Placebo into the intranasal mucosa; Drug: 20 IU NovoLog Insulin aspart into the intranasal mucosa; Drug: 40 IU NovoLog Insulin aspart into the intranasal mucosa; Drug: 60 IU NovoLog Insulin aspart into the intranasal mucosa; Drug: 80 IU NovoLog Insulin aspart into the intranasal mucosa; Drug: 100 IU NovoLog Insulin aspart into the intranasal mucosa; Drug: 120 IU NovoLog Insulin aspart into the intranasal mucosa

INTERVENTIONS:
Drug: Placebo into the intranasal mucosa — 6 doses of 0.2mL saline solution administered into the intranasal mucosa using the MAD Nasal Atomizer
  Other Names: Saline
Drug: 20 IU NovoLog Insulin aspart into the intranasal mucosa — 5 doses of 0.2mL saline solution, 1 dose of 0.2mL NovoLog Insulin aspart (20 IU) administered into the intranasal mucosa using the MAD Nasal Atomizer
  Other Names: NovoLog Insulin aspart
Drug: 40 IU NovoLog Insulin aspart into the intranasal mucosa — 4 doses of 0.2mL saline solution, 2 doses of 0.2mL NovoLog Insulin aspart (40 IU) administered into the intranasal mucosa using the MAD Nasal Atomizer
  Other Names: NovoLog Insulin aspart
Drug: 60 IU NovoLog Insulin aspart into the intranasal mucosa — 3 doses of 0.2mL saline solution, 3 doses of 0.2mL NovoLog Insulin aspart (60 IU) administered into the intranasal mucosa using the MAD Nasal Atomizer
  Other Names: NovoLog Insulin aspart
Drug: 80 IU NovoLog Insulin aspart into the intranasal mucosa — 2 doses of 0.2mL saline solution, 4 doses of 0.2mL NovoLog Insulin aspart (80 IU) administered into the intranasal mucosa using the MAD Nasal Atomizer
  Other Names: NovoLog Insulin aspart
Drug: 100 IU NovoLog Insulin aspart into the intranasal mucosa — 1 dose of 0.2mL saline solution, 5 doses of 0.2mL NovoLog Insulin aspart (100 IU) administered into the intranasal mucosa using the MAD Nasal Atomizer
  Other Names: NovoLog Insulin aspart
Drug: 120 IU NovoLog Insulin aspart into the intranasal mucosa — 6 doses of 0.2mL NovoLog Insulin aspart (120 IU) administered into the intranasal mucosa using the MAD Nasal Atomizer
  Other Names: NovoLog Insulin aspart

SUMMARY:
To determine if physical activity engagement alters the dose-response profile and safety of administration of insulin into the intranasal mucosa.

DETAILED DESCRIPTION:
Using a randomized placebo controlled double-blind pre-posttest design, participants will be randomly assigned to receive a dose of either 0, 20, 40, 60, 80, 100, or 120 IU of NovoLog insulin aspart prior to being randomized into participating in a 20 minute session of either moderate-intensity aerobic exercise or a passive control condition. The efficacy of the intranasal insulin for inducing alterations in cognition will be assessed using both behavioral and neuroelectric measures. The safety of the protocol will be assessed using a symptom questionnaire assessing common symptoms of altered blood glucose and common side effects of intranasal insulin.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be over the age of 18..
2. Participants must have normal or corrected-to-normal vision in order to complete the cognitive task.

Exclusion Criteria:

1. Lack of consent.
2. Presence of any major neurological health issues, brain trauma, or concussion with loss of consciousness assessed through a health history and demographics questionnaire.
3. Type I or Type II Diabetes
4. Self-reported pregnancy
5. Currently has any type of inflammation or blockage of the nasal passageways (i.e. allergies or a cold affecting the sinuses).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew B Pontifex, Ph.D., Principal Investigator — Michigan State University
Locations (1):
- Department of Kinesiology, East Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will be by request and approval of the Michigan State University Human Research Protections Program with the provision of a data-safety and sharing agreement. No individually identifiable information will be shared.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available following primary publication of the results.
Access Criteria: By request

REFERENCES:
- [Derived] Gwizdala KL, Ferguson DP, Kovan J, Novak V, Pontifex MB. Placebo controlled phase II clinical trial: Safety and efficacy of combining intranasal insulin & acute exercise. Metab Brain Dis. 2021 Aug;36(6):1289-1303. doi: 10.1007/s11011-021-00727-2. Epub 2021 Apr 15. PMID 33856613

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the mid-Michigan area.
Pre-assignment Details: 177 individuals were assessed for eligibility. 61 individuals were excluded (58 for failing medical screening, 1 diabetic, 1 unable to exercise, 1 history of epilepsy) 116 individuals were randomized using a serial stratification approach.
Groups:
- Passive Control - Placebo: 20 minute sedentary control period during which participants watched an emotionally neutral video.
  Placebo into the intranasal mucosa: 6 doses of 0.2mL saline solution administered into the intranasal mucosa using the MAD Nasal Atomizer
- Passive Control - 20 IU: 20 minute sedentary control period during which participants watched an emotionally neutral video.
  20 IU NovoLog Insulin aspart into the intranasal mucosa: 5 doses of 0.2mL saline solution, 1 dose of 0.2mL NovoLog Insulin aspart (20 IU) administered into the intranasal mucosa using the MAD Nasal Atomizer
- Passive Control - 40 IU: 20 minute sedentary control period during which participants watched an emotionally neutral video.
  40 IU NovoLog Insulin aspart into the intranasal mucosa: 4 doses of 0.2mL saline solution, 2 doses of 0.2mL NovoLog Insulin aspart (40 IU) administered into the intranasal mucosa using the MAD Nasal Atomizer
- Passive Control - 60 IU: 20 minute sedentary control period during which participants watched an emotionally neutral video.
  60 IU NovoLog Insulin aspart into the intranasal mucosa: 3 doses of 0.2mL saline solution, 3 doses of 0.2mL NovoLog Insulin aspart (60 IU) administered into the intranasal mucosa using the MAD Nasal Atomizer
- Passive Control - 80 IU: 20 minute sedentary control period during which participants watched an emotionally neutral video.
  80 IU NovoLog Insulin aspart into the intranasal mucosa: 2 doses of 0.2mL saline solution, 4 doses of 0.2mL NovoLog Insulin aspart (80 IU) administered into the intranasal mucosa using the MAD Nasal Atomizer
- Passive Control - 100 IU: 20 minute sedentary control period during which participants watched an emotionally neutral video.
  100 IU NovoLog Insulin aspart into the intranasal mucosa: 1 dose of 0.2mL saline solution, 5 doses of 0.2mL NovoLog Insulin aspart (100 IU) administered into the intranasal mucosa using the MAD Nasal Atomizer
- Passive Control - 120 IU: 20 minute sedentary control period during which participants watched an emotionally neutral video.
  120 IU NovoLog Insulin aspart into the intranasal mucosa: 6 doses of 0.2mL NovoLog Insulin aspart (120 IU) administered into the intranasal mucosa using the MAD Nasal Atomizer
- Acute Exercise - Placebo: 20 minute physical activity period during which participants exercised on a treadmill at 60-65% of maximum heart rate.
  Placebo into the intranasal mucosa: 6 doses of 0.2mL saline solution administered into the intranasal mucosa using the MAD Nasal Atomizer
- Acute Exercise - 20 IU: 20 minute physical activity period during which participants exercised on a treadmill at 60-65% of maximum heart rate.
  20 IU NovoLog Insulin aspart into the intranasal mucosa: 5 doses of 0.2mL saline solution, 1 dose of 0.2mL NovoLog Insulin aspart (20 IU) administered into the intranasal mucosa using the MAD Nasal Atomizer
- Acute Exercise - 40 IU: 20 minute physical activity period during which participants exercised on a treadmill at 60-65% of maximum heart rate.
  40 IU NovoLog Insulin aspart into the intranasal mucosa: 4 doses of 0.2mL saline solution, 2 doses of 0.2mL NovoLog Insulin aspart (40 IU) administered into the intranasal mucosa using the MAD Nasal Atomizer
- Acute Exercise - 60 IU: 20 minute physical activity period during which participants exercised on a treadmill at 60-65% of maximum heart rate.
  60 IU NovoLog Insulin aspart into the intranasal mucosa: 3 doses of 0.2mL saline solution, 3 doses of 0.2mL NovoLog Insulin aspart (60 IU) administered into the intranasal mucosa using the MAD Nasal Atomizer
- Acute Exercise - 80 IU: 20 minute physical activity period during which participants exercised on a treadmill at 60-65% of maximum heart rate.
  80 IU NovoLog Insulin aspart into the intranasal mucosa: 2 doses of 0.2mL saline solution, 4 doses of 0.2mL NovoLog Insulin aspart (80 IU) administered into the intranasal mucosa using the MAD Nasal Atomizer
- Acute Exercise - 100 IU: 20 minute physical activity period during which participants exercised on a treadmill at 60-65% of maximum heart rate.
  100 IU NovoLog Insulin aspart into the intranasal mucosa: 1 dose of 0.2mL saline solution, 5 doses of 0.2mL NovoLog Insulin aspart (100 IU) administered into the intranasal mucosa using the MAD Nasal Atomizer
- Acute Exercise - 120 IU: 20 minute physical activity period during which participants exercised on a treadmill at 60-65% of maximum heart rate.
  120 IU NovoLog Insulin aspart into the intranasal mucosa: 6 doses of 0.2mL NovoLog Insulin aspart (120 IU) administered into the intranasal mucosa using the MAD Nasal Atomizer
Period: Overall Study
Arm/Group | Passive Control - Placebo | Passive Control - 20 IU | Passive Control - 40 IU | Passive Control - 60 IU | Passive Control - 80 IU | Passive Control - 100 IU | Passive Control - 120 IU | Acute Exercise - Placebo | Acute Exercise - 20 IU | Acute Exercise - 40 IU | Acute Exercise - 60 IU | Acute Exercise - 80 IU | Acute Exercise - 100 IU | Acute Exercise - 120 IU
Started | 8 | 8 | 9 | 8 | 8 | 9 | 8 | 10 | 8 | 8 | 7 | 7 | 9 | 9
Completed | 8 | 8 | 9 | 8 | 8 | 9 | 8 | 8 (Condition stopped due to Blood Sugar Below 70 mg/dL (n = 1)) | 8 | 8 | 7 | 6 | 8 (Condition stopped due to Blood Sugar Below 70 mg/dL (n = 1)) | 7 (Condition stopped due to Blood Sugar Below 70 mg/dL (n = 1) Condition stopped due to Report of Dizziness (n = 1))
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Condition stopped due to Blood Sugar Below 70 mg/dL | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Report of Dizziness | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Equipment Failure | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Passive Control - Placebo | Passive Control - 20 IU | Passive Control - 40 IU | Passive Control - 60 IU | Passive Control - 80 IU | Passive Control - 100 IU | Passive Control - 120 IU | Acute Exercise - Placebo | Acute Exercise - 20 IU | Acute Exercise - 40 IU | Acute Exercise - 60 IU | Acute Exercise - 80 IU | Acute Exercise - 100 IU | Acute Exercise - 120 IU | Total
Number analyzed (Participants) | 8 | 8 | 9 | 8 | 8 | 9 | 8 | 10 | 8 | 8 | 7 | 7 | 9 | 9 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.8 (2.0) | 20.7 (1.4) | 20.0 (0.9) | 21.9 (3.1) | 19.6 (1.3) | 20.8 (2.5) | 23.1 (3.9) | 19.8 (1.5) | 19.9 (1.5) | 21.8 (3.9) | 21.3 (3.9) | 20.2 (1.8) | 20.1 (1.4) | 20.1 (2.4) | 20.7 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 6 | 5 | 5 | 6 | 5 | 6 | 5 | 5 | 4 | 4 | 6 | 5 | 72
  Male | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 4 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 7
  Not Hispanic or Latino | 8 | 6 | 8 | 8 | 7 | 8 | 7 | 10 | 8 | 7 | 7 | 7 | 9 | 9 | 109
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3
  White | 7 | 7 | 8 | 5 | 6 | 9 | 6 | 8 | 6 | 6 | 5 | 6 | 9 | 8 | 96
  More than one race | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 8 | 9 | 8 | 8 | 9 | 8 | 10 | 8 | 8 | 7 | 7 | 9 | 9 | 116
Education [Mean (Standard Deviation); unit: years] | 14.4 (1.9) | 14.2 (1.3) | 13.7 (1.2) | 14.4 (2.8) | 13.6 (2.7) | 13.4 (2.3) | 15.6 (2.6) | 13.0 (1.1) | 13.2 (1.9) | 15.1 (3.4) | 14.0 (2.8) | 13.7 (2.1) | 13.4 (1.4) | 13.2 (1.9) | 13.9 (2.2)
WASI-II (IQ) [Mean (Standard Deviation); unit: units on a scale] — Wechsler Abbreviated Scale of Intelligence (2nd Edition) Scores represents performance on the Vocabulary and Matrix Reasoning subtests. For each test the scores are converted to T scores. T scores on each scale are summed together. Scores range from 45 to 160 with higher values representing better performance.
  units on a scale | 104.7 (6.6) | 105.0 (7.6) | 98.3 (8.1) | 110.0 (6.4) | 113.6 (10.1) | 120.6 (12.7) | 110.7 (10.5) | 104.4 (4.3) | 110.8 (18.8) | 107.7 (8.0) | 110.8 (4.1) | 103.5 (8.7) | 108.2 (16.8) | 101.2 (17.8) | 107.5 (9.9)
Fasting blood glucose (mg/dL) [Mean (Standard Deviation); unit: mg/dL] | 94.1 (6.9) | 96.0 (10.3) | 99.0 (9.3) | 91.9 (3.5) | 96.4 (6.5) | 94.4 (9.4) | 97.8 (7.3) | 92.2 (9.4) | 97.4 (7.9) | 87.1 (9.6) | 93.1 (9.3) | 96.3 (7.3) | 92.7 (9.6) | 96.0 (9.5) | 94.6 (8.6)
Aerobic fitness percentile [Mean (Standard Deviation); unit: percentile] — Relative peak oxygen consumption (ml/kg/min) was measured using indirect calorimetry during a maximal exercise test and then converted to percentiles based upon normative data taking into account age and biological sex. Percentiles range from 3 to 97 with higher values reflecting a greater aerobic capacity.
  percentile | 44.7 (28.8) | 26.2 (10.7) | 68.5 (12.9) | 54.5 (24.0) | 35.9 (23.1) | 53.6 (36.3) | 41.7 (26.9) | 59.2 (26.9) | 45.2 (23.7) | 48.7 (34.5) | 52.0 (28.5) | 55.8 (23.2) | 71.8 (23.2) | 28.8 (10.0) | 46.9 (24.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Manifestation of Any Symptom at Any Point During the Protocol
Description: The manifestation of any symptom that could be associated with alterations in blood glucose and side effects of intranasal insulin. Fewer symptoms would indicate a better outcome. Burning/tingling of the nose and watering/tearing of the eyes during the nasal spray were the most cited symptoms.
Time Frame: During the 20 minute exercise/control period and the cognitive assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Passive Control - Placebo | Passive Control - 20 IU | Passive Control - 40 IU | Passive Control - 60 IU | Passive Control - 80 IU | Passive Control - 100 IU | Passive Control - 120 IU | Acute Exercise - Placebo | Acute Exercise - 20 IU | Acute Exercise - 40 IU | Acute Exercise - 60 IU | Acute Exercise - 80 IU | Acute Exercise - 100 IU | Acute Exercise - 120 IU
Number analyzed (Participants) | 8 | 8 | 9 | 8 | 8 | 9 | 8 | 10 | 8 | 8 | 7 | 7 | 9 | 9
Participants | 4 | 6 | 6 | 4 | 5 | 9 | 5 | 2 | 4 | 3 | 4 | 4 | 7 | 9

2. Primary Outcome: Number of Participants With Manifestation of Any Symptom Following the Protocol
Description: The manifestation of any symptom that could be associated with alterations in blood glucose and side effects of intranasal insulin. Fewer symptoms would indicate a better outcome. The most cited symptom was having a runny nose.
Time Frame: Approximately 1 hour following the dose of intranasal insulin (~32 minutes following the end of the passive control/exercise condition; immediately following the completion of the post-test cognitive assessments)
Measure: Count of Participants; unit: Participants
Arm/Group | Passive Control - Placebo | Passive Control - 20 IU | Passive Control - 40 IU | Passive Control - 60 IU | Passive Control - 80 IU | Passive Control - 100 IU | Passive Control - 120 IU | Acute Exercise - Placebo | Acute Exercise - 20 IU | Acute Exercise - 40 IU | Acute Exercise - 60 IU | Acute Exercise - 80 IU | Acute Exercise - 100 IU | Acute Exercise - 120 IU
Number analyzed (Participants) | 8 | 8 | 9 | 8 | 8 | 9 | 8 | 10 | 8 | 8 | 7 | 7 | 9 | 9
Participants | 1 | 2 | 0 | 2 | 1 | 4 | 3 | 0 | 1 | 2 | 1 | 0 | 3 | 2

3. Primary Outcome: Effect Size for Change in Behavioral Index of Inhibitory Control - RT
Description: The effect size of the change from pre-to-posttest in behavioral metrics of performance (RT) on a flanker test of inhibitory control. A more negative effect size would indicate a better outcome. Effect sizes were computed for each participant as the standardized change relative to the pretest assessment using the within-subject (drm) variance correction for Cohen's d (Lakens, 2013). To ensure the integrity of the effect size estimates, within-subject effect sizes exceeding 3 times the interquartile range were identified as outliers and removed from analysis.
  Effect sizes are computed per Arm and do not reflect comparisons or combinations across Arms/Groups.
Time Frame: Prior to intranasal insulin administration relative to 30 minutes following
Measure: Mean (95% Confidence Interval); unit: cohens d
Arm/Group | Passive Control - Placebo | Passive Control - 20 IU | Passive Control - 40 IU | Passive Control - 60 IU | Passive Control - 80 IU | Passive Control - 100 IU | Passive Control - 120 IU | Acute Exercise - Placebo | Acute Exercise - 20 IU | Acute Exercise - 40 IU | Acute Exercise - 60 IU | Acute Exercise - 80 IU | Acute Exercise - 100 IU | Acute Exercise - 120 IU
Number analyzed (Participants) | 8 | 8 | 9 | 8 | 8 | 9 | 8 | 8 | 8 | 8 | 7 | 7 | 8 | 7
cohens d | -0.04 [-0.17 to 0.09] | -0.29 [-0.45 to -0.13] | -0.54 [-0.81 to -0.27] | -0.10 [-0.38 to 0.18] | -0.42 [-0.61 to -0.23] | -0.25 [-0.54 to -0.03] | -0.10 [-0.29 to 0.09] | -0.08 [-0.26 to 0.10] | -0.20 [-0.40 to 0.01] | -0.25 [-0.42 to -0.08] | -0.33 [-0.63 to -0.04] | -0.19 [-0.42 to 0.04] | -0.27 [-0.57 to 0.03] | -0.36 [-0.55 to -0.16]

4. Primary Outcome: Effect Size for Change in Behavioral Index of Inhibitory Control - Accuracy
Description: The effect size of the change from pre-to-posttest in behavioral metrics of performance (response accuracy) on a flanker test of inhibitory control. A more positive effect size would indicate a better outcome. Effect sizes were computed for each participant as the standardized change relative to the pretest assessment using the within-subject (drm) variance correction for Cohen's d (Lakens, 2013). To ensure the integrity of the effect size estimates, within-subject effect sizes exceeding 3 times the interquartile range were identified as outliers and removed from analysis.
  Effect sizes are computed per Arm and do not reflect comparisons or combinations across Arms/Groups.
Time Frame: Prior to intranasal insulin administration relative to 30 minutes following
Measure: Mean (95% Confidence Interval); unit: cohens d
Arm/Group | Passive Control - Placebo | Passive Control - 20 IU | Passive Control - 40 IU | Passive Control - 60 IU | Passive Control - 80 IU | Passive Control - 100 IU | Passive Control - 120 IU | Acute Exercise - Placebo | Acute Exercise - 20 IU | Acute Exercise - 40 IU | Acute Exercise - 60 IU | Acute Exercise - 80 IU | Acute Exercise - 100 IU | Acute Exercise - 120 IU
Number analyzed (Participants) | 8 | 8 | 9 | 8 | 8 | 9 | 8 | 8 | 8 | 8 | 7 | 7 | 8 | 7
cohens d | -0.03 [-0.28 to 0.22] | 0.16 [-0.17 to 0.49] | -0.04 [-0.28 to 0.21] | -0.19 [-0.40 to 0.02] | -0.06 [-0.37 to 0.26] | -0.14 [-0.46 to 0.19] | -0.05 [-0.14 to 0.05] | 0.05 [-0.23 to 0.33] | -0.26 [-0.74 to 0.23] | -0.12 [-0.51 to 0.28] | 0.06 [-0.18 to 0.29] | -0.01 [-0.25 to 0.23] | 0.01 [-0.26 to 0.27] | -0.13 [-0.46 to 0.20]

5. Primary Outcome: Effect Size of Change in Neuroelectric Index of Attentional Engagement - Inhibition Task
Description: The effect size of the change from pre-to-posttest in neuroelectric measures of attention (P3b amplitude) in response to the flanker test of inhibitory control. The effect size was collapsed across a nine-channel region-of-interest centering around the topographic maxima of the P3 (i.e., the CP3/Z/4, P3/Z/4, PO5/Z/6 electrodes). A larger effect size would indicate a better outcome. Effect sizes were computed for each participant as the standardized change relative to the pretest assessment using the within-subject (drm) variance correction for Cohen's d (Lakens, 2013). To ensure the integrity of the effect size estimates, within-subject effect sizes exceeding 3 times the interquartile range were identified as outliers and removed from analysis.
  Effect sizes are computed per Arm and do not reflect comparisons or combinations across Arms/Groups.
Time Frame: Prior to intranasal insulin administration relative to 30 minutes following
Measure: Mean (95% Confidence Interval); unit: cohens d
Arm/Group | Passive Control - Placebo | Passive Control - 20 IU | Passive Control - 40 IU | Passive Control - 60 IU | Passive Control - 80 IU | Passive Control - 100 IU | Passive Control - 120 IU | Acute Exercise - Placebo | Acute Exercise - 20 IU | Acute Exercise - 40 IU | Acute Exercise - 60 IU | Acute Exercise - 80 IU | Acute Exercise - 100 IU | Acute Exercise - 120 IU
Number analyzed (Participants) | 8 | 8 | 9 | 8 | 8 | 9 | 8 | 8 | 8 | 8 | 7 | 6 | 8 | 7
cohens d | 0.07 [-0.04 to 0.17] | -0.08 [-0.24 to 0.08] | -0.01 [-0.12 to 0.10] | 0.00 [-0.09 to 0.08] | 0.00 [-0.15 to 0.15] | -0.06 [-0.20 to 0.07] | 0.00 [-0.12 to 0.12] | 0.00 [-0.09 to 0.09] | 0.00 [-0.08 to 0.08] | -0.04 [-0.16 to 0.09] | 0.01 [-0.17 to 0.19] | -0.03 [-0.11 to 0.04] | 0.00 [-0.09 to 0.10] | 0.15 [0.09 to 0.21]

6. Primary Outcome: Effect Size of Change in Neuroelectric Index of Attentional Processing Speed - Inhibition Task
Description: The effect size of the change from pre-to-posttest in neuroelectric measures of attention (P3b latency) in response to the flanker test of inhibitory control. The effect size was collapsed across a nine-channel region-of-interest centering around the topographic maxima of the P3 (i.e., the CP3/Z/4, P3/Z/4, PO5/Z/6 electrodes). A smaller effect size would indicate a better outcome. Effect sizes were computed for each participant as the standardized change relative to the pretest assessment using the within-subject (drm) variance correction for Cohen's d (Lakens, 2013). To ensure the integrity of the effect size estimates, within-subject effect sizes exceeding 3 times the interquartile range were identified as outliers and removed from analysis.
  Effect sizes are computed per Arm and do not reflect comparisons or combinations across Arms/Groups.
Time Frame: Prior to intranasal insulin administration relative to 30 minutes following
Measure: Mean (95% Confidence Interval); unit: cohens d
Arm/Group | Passive Control - Placebo | Passive Control - 20 IU | Passive Control - 40 IU | Passive Control - 60 IU | Passive Control - 80 IU | Passive Control - 100 IU | Passive Control - 120 IU | Acute Exercise - Placebo | Acute Exercise - 20 IU | Acute Exercise - 40 IU | Acute Exercise - 60 IU | Acute Exercise - 80 IU | Acute Exercise - 100 IU | Acute Exercise - 120 IU
Number analyzed (Participants) | 8 | 8 | 9 | 8 | 8 | 9 | 8 | 8 | 8 | 8 | 7 | 6 | 8 | 7
cohens d | -0.22 [-0.54 to 0.10] | -0.06 [-0.30 to 0.19] | 0.16 [-0.14 to 0.45] | 0.15 [-0.28 to 0.58] | -0.42 [-1.00 to 0.16] | 0.06 [-0.14 to 0.26] | -0.05 [-0.53 to 0.42] | -0.21 [-0.40 to -0.03] | -0.03 [-0.37 to 0.31] | -0.25 [-0.52 to 0.02] | -0.41 [-0.98 to 0.16] | 0.12 [-0.40 to 0.64] | 0.19 [-0.54 to 0.93] | 0.20 [-0.35 to 0.75]

7. Primary Outcome: Effect Size of Change in Behavioral Index of Sustained Attention - RT
Description: The effect size of the change from pre-to-posttest in behavioral metrics of performance (RT) on a Rapid Visual Information Processing test of sustained attention. A more negative effect size would indicate a better outcome. Effect sizes were computed for each participant as the standardized change relative to the pretest assessment using the within-subject (drm) variance correction for Cohen's d (Lakens, 2013). To ensure the integrity of the effect size estimates, within-subject effect sizes exceeding 3 times the interquartile range were identified as outliers and removed from analysis.
  Effect sizes are computed per Arm and do not reflect comparisons or combinations across Arms/Groups.
Time Frame: Prior to intranasal insulin administration relative to 30 minutes following
Measure: Mean (95% Confidence Interval); unit: cohens d
Arm/Group | Passive Control - Placebo | Passive Control - 20 IU | Passive Control - 40 IU | Passive Control - 60 IU | Passive Control - 80 IU | Passive Control - 100 IU | Passive Control - 120 IU | Acute Exercise - Placebo | Acute Exercise - 20 IU | Acute Exercise - 40 IU | Acute Exercise - 60 IU | Acute Exercise - 80 IU | Acute Exercise - 100 IU | Acute Exercise - 120 IU
Number analyzed (Participants) | 8 | 8 | 9 | 8 | 8 | 9 | 8 | 8 | 8 | 8 | 7 | 7 | 8 | 7
cohens d | -0.18 [-0.37 to 0.00] | -0.16 [-0.25 to -0.07] | -0.15 [-0.49 to 0.19] | -0.24 [-0.54 to 0.06] | -0.20 [-0.36 to -0.03] | -0.22 [-0.37 to -0.07] | -0.11 [-0.37 to 0.15] | -0.16 [-0.29 to -0.03] | -0.05 [-0.16 to 0.07] | -0.16 [-0.54 to 0.23] | -0.18 [-0.36 to 0.01] | -0.09 [-0.26 to 0.09] | -0.19 [-0.39 to 0.00] | -0.16 [-0.37 to 0.06]

8. Primary Outcome: Effect Size of Change in Behavioral Index of Sustained Attention - Accuracy
Description: The effect size of the change from pre-to-posttest in behavioral metrics of performance (response accuracy) on a Rapid Visual Information Processing test of sustained attention. A more positive effect size would indicate a better outcome. Effect sizes were computed for each participant as the standardized change relative to the pretest assessment using the within-subject (drm) variance correction for Cohen's d (Lakens, 2013). To ensure the integrity of the effect size estimates, within-subject effect sizes exceeding 3 times the interquartile range were identified as outliers and removed from analysis.
  Effect sizes are computed per Arm and do not reflect comparisons or combinations across Arms/Groups.
Time Frame: Prior to intranasal insulin administration relative to 30 minutes following
Measure: Mean (95% Confidence Interval); unit: cohens d
Arm/Group | Passive Control - Placebo | Passive Control - 20 IU | Passive Control - 40 IU | Passive Control - 60 IU | Passive Control - 80 IU | Passive Control - 100 IU | Passive Control - 120 IU | Acute Exercise - Placebo | Acute Exercise - 20 IU | Acute Exercise - 40 IU | Acute Exercise - 60 IU | Acute Exercise - 80 IU | Acute Exercise - 100 IU | Acute Exercise - 120 IU
Number analyzed (Participants) | 8 | 8 | 9 | 8 | 8 | 9 | 8 | 8 | 8 | 8 | 7 | 7 | 8 | 7
cohens d | 0.69 [0.19 to 1.20] | 0.81 [-0.10 to 1.73] | 0.05 [-0.51 to 0.62] | 0.87 [0.40 to 1.35] | 0.62 [0.03 to 1.20] | 0.71 [0.10 to 1.32] | 0.69 [-0.13 to 1.51] | 0.54 [0.06 to 1.02] | 0.36 [-0.07 to 0.80] | -0.21 [-1.23 to 0.80] | 0.78 [0.23 to 1.32] | 0.43 [-0.12 to 0.98] | 0.90 [0.33 to 1.48] | 0.60 [-0.23 to 1.44]

9. Primary Outcome: Effect Size of Change in Neuroelectric Index of Attentional Engagement - RVIP Task
Description: The effect size of the change from pre-to-posttest in neuroelectric measures of attention (P3b amplitude) in response to the target trial of the Rapid Visual Information Processing test of sustained attention. The effect size was collapsed across a nine-channel region-of-interest centering around the topographic maxima of the P3 (i.e., the CP3/Z/4, P3/Z/4, PO5/Z/6 electrodes). A larger effect size would indicate a better outcome. Effect sizes were computed for each participant as the standardized change relative to the pretest assessment using the within-subject (drm) variance correction for Cohen's d (Lakens, 2013). To ensure the integrity of the effect size estimates, within-subject effect sizes exceeding 3 times the interquartile range were identified as outliers and removed from analysis. Effect sizes are computed per Arm and do not reflect comparisons or combinations across Arms/Groups.
Time Frame: Prior to intranasal insulin administration relative to 30 minutes following
Measure: Mean (95% Confidence Interval); unit: cohens d
Arm/Group | Passive Control - Placebo | Passive Control - 20 IU | Passive Control - 40 IU | Passive Control - 60 IU | Passive Control - 80 IU | Passive Control - 100 IU | Passive Control - 120 IU | Acute Exercise - Placebo | Acute Exercise - 20 IU | Acute Exercise - 40 IU | Acute Exercise - 60 IU | Acute Exercise - 80 IU | Acute Exercise - 100 IU | Acute Exercise - 120 IU
Number analyzed (Participants) | 8 | 8 | 9 | 8 | 8 | 9 | 8 | 8 | 8 | 8 | 7 | 6 | 8 | 7
cohens d | -0.02 [-0.27 to 0.23] | -0.09 [-0.21 to 0.03] | 0.04 [-0.20 to 0.29] | 0.23 [0.02 to 0.45] | 0.02 [-0.17 to 0.21] | 0.16 [0.03 to 0.28] | 0.08 [-0.15 to 0.31] | 0.03 [-0.17 to 0.24] | 0.02 [-0.18 to 0.22] | 0.02 [-0.15 to 0.20] | 0.18 [0.00 to 0.36] | 0.04 [-0.25 to 0.33] | -0.03 [-0.19 to 0.14] | -0.06 [-0.35 to 0.24]

10. Primary Outcome: Effect Size of Change in Neuroelectric Index of Attentional Processing Speed - RVIP Task
Description: The effect size of the change from pre-to-posttest in neuroelectric measures of attention (P3b latency) in response to the target trial of the Rapid Visual Information Processing test of sustained attention. The effect size was collapsed across a nine-channel region-of-interest centering around the topographic maxima of the P3 (i.e., the CP3/Z/4, P3/Z/4, PO5/Z/6 electrodes). A smaller effect size would indicate a better outcome. Effect sizes were computed for each participant as the standardized change relative to the pretest assessment using the within-subject (drm) variance correction for Cohen's d (Lakens, 2013). To ensure the integrity of the effect size estimates, within-subject effect sizes exceeding 3 times the interquartile range were identified as outliers and removed from analysis.
  Effect sizes are computed per Arm and do not reflect comparisons or combinations across Arms/Groups.
Time Frame: Prior to intranasal insulin administration relative to 30 minutes following
Measure: Mean (95% Confidence Interval); unit: cohens d
Arm/Group | Passive Control - Placebo | Passive Control - 20 IU | Passive Control - 40 IU | Passive Control - 60 IU | Passive Control - 80 IU | Passive Control - 100 IU | Passive Control - 120 IU | Acute Exercise - Placebo | Acute Exercise - 20 IU | Acute Exercise - 40 IU | Acute Exercise - 60 IU | Acute Exercise - 80 IU | Acute Exercise - 100 IU | Acute Exercise - 120 IU
Number analyzed (Participants) | 8 | 8 | 9 | 8 | 8 | 9 | 8 | 8 | 8 | 8 | 7 | 6 | 8 | 7
cohens d | 0.08 [-0.32 to 0.48] | -0.06 [-0.26 to 0.14] | -0.08 [-0.77 to 0.61] | -0.09 [-0.29 to 0.11] | 0.26 [-0.43 to 0.96] | 0.25 [-0.36 to 0.86] | -0.10 [-0.48 to 0.29] | -0.03 [-0.33 to 0.27] | 0.34 [-0.15 to 0.83] | 0.00 [-0.22 to 0.21] | 0.04 [-0.30 to 0.37] | 0.05 [-0.30 to 0.40] | 0.10 [-0.36 to 0.57] | 0.05 [-0.37 to 0.47]

ADVERSE EVENTS:
Time Frame: Only during the two 90 minute sessions.
Description: The clinicaltrials.gov definitions for adverse events was used. Indications of onset of an issue related to hypoglycemia were stopping criteria for the study protocol and are considered herein as Non serious adverse events.
Arm/Group | Passive Control - Placebo | Passive Control - 20 IU | Passive Control - 40 IU | Passive Control - 60 IU | Passive Control - 80 IU | Passive Control - 100 IU | Passive Control - 120 IU | Acute Exercise - Placebo | Acute Exercise - 20 IU | Acute Exercise - 40 IU | Acute Exercise - 60 IU | Acute Exercise - 80 IU | Acute Exercise - 100 IU | Acute Exercise - 120 IU
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/9 | 0/8 | 0/8 | 0/9 | 0/8 | 0/10 | 0/8 | 0/8 | 0/7 | 0/7 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/9 | 0/8 | 0/8 | 0/9 | 0/8 | 0/10 | 0/8 | 0/8 | 0/7 | 0/7 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/9 | 0/8 | 0/8 | 0/9 | 0/8 | 1/10 | 0/8 | 0/8 | 0/7 | 0/7 | 1/9 | 2/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Passive Control - Placebo (N=8) | Passive Control - 20 IU (N=8) | Passive Control - 40 IU (N=9) | Passive Control - 60 IU (N=8) | Passive Control - 80 IU (N=8) | Passive Control - 100 IU (N=9) | Passive Control - 120 IU (N=8) | Acute Exercise - Placebo (N=10) | Acute Exercise - 20 IU (N=8) | Acute Exercise - 40 IU (N=8) | Acute Exercise - 60 IU (N=7) | Acute Exercise - 80 IU (N=7) | Acute Exercise - 100 IU (N=9) | Acute Exercise - 120 IU (N=9)
Hypoglycemic event (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) — Blood sugar fell below 70 mg/Dl or exhibited Dizziness

LIMITATIONS AND CAVEATS:
As the present investigation was a Phase II Clinical Trial, the research design was not sufficiently powered for hypothesis testing. Given the potential risk of combining exercise with intranasal insulin the present investigation utilized a sample of healthy, non-diabetic, fasted college-aged adults to limit the potential for a serious adverse event.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/35/NCT04292535/Prot_SAP_000.pdf